CLINICAL TRIAL: NCT05437510
Title: A Phase IIIb Randomized Open-label Study of Nirsevimab (Versus no Intervention) in Preventing Hospitalizations Due to Respiratory Syncytial Virus in Infants (HARMONIE)
Brief Title: Study of a Single Intramuscular Dose of Nirsevimab in the Prevention of Hospitalizations Due to Respiratory Syncytial Virus (RSV) Infection in Healthy Term and Preterm Infants During the First Year of Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAS00006; U1111-1272-2514 (Registry Identifier: ICTRP); 2022-000099-20 (EudraCT Number)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: RSV Immunization; Healthy Volunteer
MeSH Terms: interventions — nirsevimab

STUDY DESIGN:
Intervention Model Description: 1 in-person randomization visit, with monthly safety and efficacy follow-up conducted through electronic contact through the first 6 months post-dosing/randomization.
  The study also included a 12-month (D366) follow-up telephone call. The D366 follow-up telephone call was the final follow-up telephone call for France, Germany and UK non-reconsented participants. The study included an 18-month (D546) and a 24-month (D731, final telephone call) follow-up telephone call for UK reconsented participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nirsevimab (Experimental): 1 intramuscular injection at Day 01
  Interventions: Biological: Nirsevimab
- No preventive intervention for RSV (No Intervention): No intervention

INTERVENTIONS:
Biological: Nirsevimab — Pharmaceutical Form: Solution for Injection Route of Administration: Intramuscular
  Arms: Nirsevimab

SUMMARY:
The purpose of this study was to determine the efficacy and safety of a single intramuscular (IM) dose of nirsevimab, compared to no intervention, for the prevention of hospitalizations due to lower respiratory tract infection (LRTI) caused by confirmed RSV infection (henceforth referred to as RSV LRTI hospitalizations) in all infants under 12 months of age who were not eligible to receive palivizumab.

The visit frequency was 1 in-person dosing/randomization visit, with monthly safety follow-up electronic contacts through the first 6 months post dosing/randomization for all participants. The study also included a 12-month (Day 366) follow-up telephone call. The D366 follow-up telephone call was the final follow-up telephone call for France, Germany and UK non-reconsented participants. The study included an 18-month (D546) and a 24-month (D731, final telephone call) follow-up telephone call for UK reconsented participants.

DETAILED DESCRIPTION:
12 months post-dosing/randomization for France, Germany and UK non-reconsented participants, 24 months post-dosing/randomization for UK reconsented participants. D01 was the day of randomization (both study groups) and immunization (nirsevimab group).

ELIGIBILITY:
Inclusion Criteria:

* Born at ≥ 29 weeks gestational age and aged 0 to 12 months (calendar age), who entered their first RSV season on the day of inclusion in the study (D01)
* Informed consent form was signed and dated by the parent(s) or other LAR(s) (and by an independent witness if required by local regulations)
* Participant and parent/LAR were able to attend the scheduled visit and to comply with all study procedures

Exclusion Criteria:

* Participants were not eligible for the study if any of the following criteria are met:
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Active confirmed RSV infection at the time of dosing/randomization
* Active LRTI at the time of dosing/randomization
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the study intervention used in the study or to a product containing any of the same substances
* Laboratory confirmed thrombocytopenia, or known thrombocytopenia, as reported by the parent/LAR, contraindicating intramuscular injection
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular injection
* Any condition that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention administration.
* A prospective participant was not included in the study until the condition has resolved or the febrile event has subsided
* Mother of the infant participant was administered an RSV vaccine during her pregnancy with the infant participant
* Receipt of any monoclonal antibody by the infant participant
* Receipt of immune globulins, blood or blood-derived products in the past 3 months by the infant participant
* Participation at the time of study enrollment or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Eligible to receive palivizumab at time of inclusion (as per local guidelines)
* In an emergency setting or hospitalized involuntarily
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study

The above information were not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8057 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2025-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (240):
- France (66):
  - Investigational Site 2500041, Aix-en-Provence
  - Investigational Site 2500002, Amiens
  - Investigational Site Number: 2500014, Bordeaux
  - Investigational Site 2500007, Brest
  - Investigational Site Number: 2500038, Brest
  - Investigational Site Number: 2500045, Brest
  - Investigational Site Number: 2500019, Bron
  - Investigational Site Number: 2500043, Brumath
  - Investigational Site Number: 2500001, Caen
  - Investigational Site Number: 2500032, Chambéry
  - Investigational Site Number: 2500057, Clamart
  - Investigational Site Number: 2500065, Clamart
  - Investigational Site Number: 2500029, Combs-la-Ville
  - Investigational Site Number: 2500013, Corbeil-Essonnes
  - Investigational Site Number: 2500054, Creil
  - Investigational Site Number: 2500006, Créteil
  - Investigational Site Number: 2500039, Créteil
  - Investigational Site Number: 2500023, Dijon
  - Investigational Site Number: 2500069, Draguignan
  - Investigational Site 2500008, Essey-lès-Nancy
  - Investigational Site 2500030, Étampes
  - Investigational Site Number: 2500058, Frouard
  - Investigational Site Number: 2500064, Grasse
  - Investigational Site Number: 2500004, Grenoble
  - Investigational Site Number: 2500027, Héry-sur-Alby
  - Investigational Site Number: 2500060, Huningue
  - Investigational Site 2500059, La Garenne-Colombes
  - Investigational Site Number: 2500071, La Teste-de-Buch
  - Investigational Site Number: 2500034, Le Kremlin-Bicêtre
  - Investigational Site Number: 2500072, Libourne
  - Investigational Site 2500046, Lille
  - Investigational Site 2500005, Lille
  - Investigational Site Number: 2500012, Limoges
  - Investigational Site Number: 2500037, Longjumeau
  - Investigational Site 2500021, Maromme
  - Investigational Site Number: 2500003, Marseille
  - Investigational Site Number: 2500073, Marseille
  - Investigational Site Number: 2500068, Mont-de-Marsan
  - Investigational Site Number: 2500066, Mont-Saint-Aignan
  - Investigational Site Number: 2500067, Montpellier
  - Investigational Site Number: 2500077, Morlaix
  - Investigational Site Number: 2500047, Nantes
  - Investigational Site Number: 2500055, Nice
  - Investigational Site Number: 2500009, Nice
  - Investigational Site Number: 2500040, Nogent-sur-Marne
  - Investigational Site Number: 2500022, Orléans
  - Investigational Site Number: 2500050, Orléans
  - Investigational Site Number: 2500024, Paris
  - Investigational Site Number: 2500010, Paris
  - Investigational Site Number: 2500075, Paris
  - Investigational Site Number: 2500051, Paris
  - Investigational Site Number:, Pau
  - Investigational Site Number: 2500018, Poissy
  - Investigational Site Number: 2500026, Puteaux
  - Investigational Site Number: 2500042, Rouen
  - Investigational Site Number: 2500078, Saint-Doulchard
  - Investigational Site Number: 2500074, Saint-Julien-en-Genevois
  - Investigational Site Number: 2500044, Saint-Maur-des-Fossés
  - Investigational Site 2500020, Saint-Sébastien-sur-Loire
  - Investigational Site Number: 2500052, Saverne
  - Investigational Site Number: 2500015, Toulouse
  - Investigational Site Number: 2500035, Tours
  - Investigational Site Number: 2500049, Vendenheim
  - Investigational Site Number: 2500011, Villeneuve-lès-Avignon
  - Investigational Site Number: 2500063, Villeneuve-Saint-Georges
  - Investigational Site 2500028, Vincennes
- Germany (66):
  - Investigational Site Number: 2760036, Augsburg
  - Investigational Site Number: 2760017, Bad Wildungen
  - Investigational Site Number: 2760099, Berlin
  - Investigational Site Number: 2760076, Berlin
  - Investigational Site Number: 2760056, Berlin
  - Investigational Site Number: 2760050, Bielefeld
  - Investigational Site Number: 2760064, Bocholt
  - Investigational Site Number: 2760098, Bochum
  - Investigational Site Number: 2760040, Bonn
  - Investigational Site Number: 2760025, Bramsche
  - Investigational Site Number: 2760018, Braunschweig
  - Investigational Site Number: 2760051, Detmold
  - Investigational Site Number: 2760085, Dortmund
  - Investigational Site Number: 2760059, Düsseldorf
  - Investigational Site Number: 2760101, Düsseldorf
  - Investigational Site Number: 2760081, Eckental
  - Investigational Site Number: 2760045, Erfurt
  - Investigational Site Number: 2760047, Forchheim
  - Investigational Site Number: 2760030, Frankfurt (Oder)
  - Investigational Site Number: 2760015, Freiburg I. Breisgau
  - Investigational Site Number: 2760079, Gera
  - Investigational Site Number: 2760005, Gilching
  - Investigational Site Number: 2760016, Göttingen
  - Investigational Site Number: 2760060, Göttingen
  - Investigational Site Number: 2760033, Hamburg
  - Investigational Site Number: 2760057, Hamburg
  - Investigational Site Number: 2760096, Hamburg
  - Investigational Site Number: 2760032, Hamm
  - Investigational Site Number: 2760007, Hanover
  - Investigational Site Number: 2760049, Heidelberg
  - Investigational Site Number: 2760008, Herford
  - Investigational Site 2760010, Hürth
  - Investigational Site Number: 2760091, Hürth
  - Investigational Site Number: 2760035, Itzehoe
  - Investigational Site Number: 2760095, Kassel
  - Investigational Site Number: 2760084, Kirchen
  - Investigational Site Number: 2760065, Krefeld
  - Investigational Site Number: 2760020, Leipzig
  - Investigational Site Number: 2760013, Leipzig
  - Investigational Site 2760006, Mainz
  - Investigational Site Number: 2760086, Mainz
  - Investigational Site Number: 2760014, Mannheim
  - Investigational Site Number: 2760023, Mönchengladbach
  - Investigational Site Number: 2760054, Mönchengladbach
  - Investigational Site Number: 2760094, München
  - Investigational Site Number: 2760034, München
  - Investigational Site Number: 2760038, München
  - Investigational Site Number: 2760019, München
  - Investigational Site Number: 2760046, München
  - Investigational Site Number: 2760061, München
  - Investigational Site Number: 2760083, Münster
  - Investigational Site Number: 2760027, Neuss
  - Investigational Site Number: 2760004, Niedernhausen
  - Investigational Site Number: 2760071, Passau
  - Investigational Site Number: 2760001, Regensburg
  - Investigational Site Number: 2760003, Rosenheim
  - Investigational Site Number: 2760062, Rüsselsheim A. Main
  - Investigational Site Number: 2760092, Saarbrücken
  - Investigational Site 2760029, Schönau
  - Investigational Site Number: 2760044, Schweigen
  - Investigational Site Number: 2760069, Suhl
  - Investigational Site Number: 2760067, Tuttlingen
  - Investigational Site Number: 2760043, Weiden
  - Investigational Site Number: 2760002, Wesel
  - Investigational Site Number: 2760093, Wolfsburg
  - Investigational Site Number: 2760028, Wolfsburg
- United Kingdom (108):
  - Investigational Site Number: 8260007, Amersham
  - Investigational Site Number: 8260096, Ashford
  - Investigational Site Number: 8260053, Banbury
  - Investigational Site Number: 8260057, Barnet
  - Investigational Site Number: 8260004, Barnsley
  - Investigational Site Number: 8260107, Basildon
  - Investigational Site Number: 8260110, Basingstoke
  - Investigational Site Number: 8260067, Bath
  - Investigational Site 8260009, Bath
  - Investigational Site Number: 8260100, Bebington
  - Investigational Site Number: 8260073, Belfast
  - Investigational Site Number: 8260095, Bicester
  - Investigational Site Number: 8260029, Blackburn
  - Investigational Site Number: 8260108, Bollington
  - Investigational Site Number: 8260085, Bolton
  - Investigational Site Number: 8260013, Bradford
  - Investigational Site Number: 8260112, Brierley Hill
  - Investigational Site Number: 8260058, Brighton
  - Investigational Site Number: 8260008, Bristol
  - Investigational Site Number: 8260019, Bristol
  - Investigational Site 8260046, Bristol
  - Investigational Site Number: 8260063, Bury St Edmunds
  - Investigational Site Number: 8260040, Cardiff
  - Investigational Site Number: 8260062, Cheltenham
  - Investigational Site Number: 8260066, Chertsey
  - Investigational Site Number: 8260061, Chippenham
  - Investigational Site Number: 8260036, Corby
  - Investigational Site Number: 8260054, Cottingham
  - Investigational Site Number: 8260035, Darlington
  - Investigational Site Number: 8260037, Darlington
  - Investigational Site Number: 8260041, Darlington
  - Investigational Site 8260064, Dorchester
  - Investigational Site Number: 8260087, Dundee
  - Investigational Site 8260018, Exeter
  - Investigational Site Number: 8260020, Gillingham
  - Investigational Site Number: 8260056, Great Yarmouth
  - Investigational Site Number: 8260069, Harrow
  - Investigational Site Number: 8260109, Highcliffe
  - Investigational Site Number: 8260101, Ipswich
  - Investigational Site Number: 8260027, Leicester
  - Investigational Site Number: 8260091, Leicester
  - Investigational Site Number: 8260074, Leicester
  - Investigational Site Number: 8260088, Liskeard
  - Investigational Site Number: 8260030, Liverpool
  - Investigational Site Number: 8260092, Liverpool
  - Investigational Site Number: 8260010, London
  - Investigational Site Number: 8260039, London
  - Investigational Site Number: 8260075, London
  - Investigational Site Number: 8260011, London
  - Investigational Site Number: 8260076, London
  - Investigational Site Number: 8260077, London
  - Investigational Site Number: 8260084, London
  - Investigational Site Number: 8260079, London
  - Investigational Site Number: 8260078, London
  - Investigational Site Number: 8260001, London
  - Investigational Site Number: 8260002, London
  - Investigational Site Number: 8260071, Macclesfield
  - Investigational Site Number: 8260015, Manchester
  - Investigational Site Number: 8260097, Margate
  - Investigational Site Number: 8260012, Middlesbrough
  - Investigational Site Number: 8260042, Milton Keynes
  - Investigational Site Number: 8260072, Nantwich
  - Investigational Site Number: 8260044, Newcastle upon Tyne
  - Investigational Site Number: 8260119, Newport
  - Investigational Site Number: 8260045, Newquay
  - Investigational Site Number: 8260024, Norwich
  - Investigational Site 8260028, Nottingham
  - Investigational Site 8260043, Nottingham
  - Investigational Site Number: 8260022, Oxford
  - Investigational Site Number: 8260003, Oxford
  - Investigational Site Number: 8260080, Penzance
  - Investigational Site Number: 8260093, Peterborough
  - Investigational Site Number: 8260081, Plymouth
  - Investigational Site Number: 8260094, Poole
  - Investigational Site 8260005, Poole
  - Investigational Site Number: 8260065, Portsmouth
  - Investigational Site Number: 8260106, Prescot
  - Investigational Site Number: 8260117, Preston
  - Investigational Site Number: 8260016, Reading
  - Investigational Site Number: 8260086, Reading
  - Investigational Site Number: 8260103, Redhill
  - Investigational Site Number: 8260105, Redruth
  - Investigational Site 8260026, Romsey
  - Investigational Site Number: 8260068, Runcorn
  - Investigational Site Number: 8260059, Salford
  - Investigational Site Number: 8260111, Salisbury
  - Investigational Site Number: 8260014, Sheffield
  - Investigational Site 8260051, Southampton
  - Investigational Site Number: 8260038, Stevenage
  - Investigational Site Number: 8260034, Stockport
  - Investigational Site Number: 8260025, Stockton-on-Tees
  - Investigational Site Number: 8260052, Sunderland
  - Investigational Site Number: 8260098, Sutton in Ashfield
  - Investigational Site Number: 8260083, Swanage
  - Investigational Site Number: 8260047, Swindon
  - Investigational Site Number: 8260115, Swinton
  - Investigational Site Number: 8260102, Tameside
  - Investigational Site Number: 8260032, Taunton
  - Investigational Site Number: 8260031, Torpoint
  - Investigational Site 8260082, Wantage
  - Investigational Site Number: 8260017, Waterlooville
  - Investigational Site Number: 8260104, Winchester
  - Investigational Site Number: 8260021, Winscombe
  - Investigational Site Number: 8260006, Witney
  - Investigational Site Number: 8260060, Witney
  - Investigational Site Number: 8260050, Yeovil
  - Investigational Site Number: 8260116, York
  - Investigational Site 8260023, York

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Munro APS, Drysdale SB, Cathie K, Flamein F, Knuf M, Collins AM, Hill HC, Kaiser F, Cohen R, Pinquier D, Vassilouthis NC, Carreno M, Moreau C, Bourron P, Marcelon L, Mari K, Roberts M, Tissieres P, Royal S, Faust SN; HARMONIE Study Group. 180-day efficacy of nirsevimab against hospitalisation for respiratory syncytial virus lower respiratory tract infections in infants (HARMONIE): a randomised, controlled, phase 3b trial. Lancet Child Adolesc Health. 2025 Jun;9(6):404-412. doi: 10.1016/S2352-4642(25)00102-6. PMID 40379431
- [Derived] Drysdale SB, Cathie K, Flamein F, Knuf M, Collins AM, Hill HC, Kaiser F, Cohen R, Pinquier D, Felter CT, Vassilouthis NC, Jin J, Bangert M, Mari K, Nteene R, Wague S, Roberts M, Tissieres P, Royal S, Faust SN; HARMONIE Study Group. Nirsevimab for Prevention of Hospitalizations Due to RSV in Infants. N Engl J Med. 2023 Dec 28;389(26):2425-2435. doi: 10.1056/NEJMoa2309189. PMID 38157500
- See also: VAS00006 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25372&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 235 investigational sites in France, Germany and the United Kingdom (UK).
Pre-assignment Details: Total 8057 participants were enrolled and randomized in 1:1 ratio to nirsevimab or no intervention group between 08 August 2022 to 28 February 2023. Participants were followed up for safety for 12-months (366 days) (for France, Germany, and UK non-reconsented participants) and for 24 months (731 days) (for UK participants who consented to take part into study extension [UK reconsented participants]). As pre-specified in protocol and SAP, results are presented by treatment group.
Groups:
- Nirsevimab: Participants received nirsevimab 50 milligrams (mg) (if weight <5 kilograms [kg]) or 100 mg (if weight ≥5 kg) as a single intramuscular (IM) injection on Day 1.
- No Intervention: Participants received no respiratory syncytial virus (RSV) preventive intervention on Day 1.
Period: Overall Study
Arm/Group | Nirsevimab | No Intervention
Started | 4038 | 4019
Randomized and Treated (1 participant of the no intervention group wrongly received the study intervention.) | 4015 | 1
Participants Entered Study Extension (UK participants who consented to take part into 12-month study extension.) | 1142 | 1084
Completed | 3747 | 3631
Not Completed | 291 | 388
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Deviation | 1 | 6
Not completed — Withdrawal by Parent/Guardian | 23 | 23
Not completed — Lost to Follow-up | 265 | 358

BASELINE CHARACTERISTICS:
Population: The All Randomized Set consisted of all participants randomly assigned to either the nirsevimab group or the no intervention group.
Groups:
- Nirsevimab: Participants received nirsevimab 50 mg (if weight <5 kg) or 100 mg (if weight ≥5 kg) as a single IM injection on Day 1.
- No Intervention: Participants received no RSV preventive intervention on Day 1.
- Total: Total of all reporting groups
Arm/Group | Nirsevimab | No Intervention | Total
Number analyzed (Participants) | 4038 | 4019 | 8057
Age, Continuous [Mean (Standard Deviation); unit: months] | 4.53 (3.342) | 4.48 (3.294) | 4.51 (3.318)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1950 | 1912 | 3862
  Male | 2088 | 2107 | 4195
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Infection (LRTI) Hospitalization Through the Respiratory Syncytial Virus Season
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths per minute (/min); 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. RSV season was the period of increased RSV infection.
Time Frame: From dosing/randomization (Day 1) up to approximately 7 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants | 11 | 64
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; The 2-sided 95% confidence interval (CI) for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 84.04, 95% CI 2-sided [69.493 to 92.411]

2. Secondary Outcome: Number of Participants With Very Severe Respiratory Syncytial Virus Lower Respiratory Tract Infection Through the Respiratory Syncytial Virus Season
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Very severe RSV LRTI was defined as RSV LRTI hospitalization with oxygen saturation <90% (at any time during hospitalization) and oxygen supplementation. Hospitalization was defined as the decision to admit to in-patient care by the treating physician. RSV season was the period of increased RSV infection.
Time Frame: From dosing/randomization (Day 1) up to approximately 7 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants | 5 | 21
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of very severe RSV LRTI in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0014, Exact method using binomial distribution; Efficacy = 77.71, 95% CI 2-sided [39.249 to 93.432]

3. Secondary Outcome: Number of Participants With Respiratory Syncytial Virus Lower Respiratory Tract Infection Hospitalization Through the Respiratory Syncytial Virus Season in Each Country
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. RSV season was the period of increased RSV infection. Number of participants with RSV LRTI hospitalization through the RSV season in France, UK, and Germany is presented.
Time Frame: From dosing/randomization (Day 1) up to approximately 7 months
Population: The All Randomized Set consisted of all participants randomly assigned to either the nirsevimab group or the no intervention group. 'Number Analyzed' indicates the number of participants with data collected for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  France: number analyzed (Participants) | 1090 | 1087
  France | 3 | 28
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 3 | 17
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 5 | 19
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The adjusted 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization. Adjustment based on Bonferroni-Holm procedure; Test type: Superiority; p < 0.0001, Exact method using binomial distribution — Adjusted p-value is reported; Efficacy = 90.70, 95% CI 2-sided [63.676 to 98.813]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The adjusted 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization. Adjustment based on Bonferroni-Holm procedure; Test type: Superiority; p = 0.0036, Exact method using binomial distribution — Adjusted p-value is reported; Efficacy = 83.20, 95% CI 2-sided [33.589 to 97.593]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The adjusted 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization. Adjustment based on Bonferroni-Holm procedure; Test type: Superiority; p = 0.0051, Exact method using binomial distribution — Adjusted p-value is reported; Efficacy = 74.62, 95% CI 2-sided [29.740 to 92.595]

4. Secondary Outcome: Number of Participants With Hospitalization for All-Cause Lower Respiratory Tract Infection Through the Respiratory Syncytial Virus Season
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. RSV season was the period of increased RSV infection. Number of participants with hospitalization for all-cause LRTI through the RSV season in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) up to approximately 7 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 48 | 106
  France: number analyzed (Participants) | 1090 | 1087
  France | 24 | 44
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 17 | 39
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 7 | 23
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of all-cause LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 57.97, 95% CI 2-sided [40.360 to 70.760]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of all-cause LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0039, Exact method using binomial distribution; Efficacy = 52.48, 95% CI 2-sided [20.121 to 72.360]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of all-cause LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0024, Exact method using binomial distribution; Efficacy = 58.62, 95% CI 2-sided [25.115 to 78.049]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of all-cause LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0037, Exact method using binomial distribution; Efficacy = 70.74, 95% CI 2-sided [29.567 to 89.396]

5. Secondary Outcome: Number of Participants With Respiratory Syncytial Virus Lower Respiratory Tract Infection Hospitalization Through 151 Days Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with RSV LRTI hospitalization through 151 days post-dosing/randomization in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) to Day 151
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 12 | 67
  France: number analyzed (Participants) | 1090 | 1087
  France | 4 | 28
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 3 | 20
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 5 | 19
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 82.44, 95% CI 2-sided [67.271 to 91.357]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 86.11, 95% CI 2-sided [60.283 to 96.459]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0004, Exact method using binomial distribution; Efficacy = 85.20, 95% CI 2-sided [50.084 to 97.183]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0055, Exact method using binomial distribution; Efficacy = 74.36, 95% CI 2-sided [29.006 to 92.518]

6. Secondary Outcome: Number of Participants With Very Severe Respiratory Syncytial Virus Lower Respiratory Tract Infection Through 151 Days Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Very severe RSV LRTI was defined as RSV LRTI hospitalization with oxygen saturation <90% (at any time during hospitalization) and oxygen supplementation. Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with very severe RSV LRTI through 151 days post-dosing/randomization in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) to Day 151
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 6 | 24
  France: number analyzed (Participants) | 1090 | 1087
  France | 2 | 9
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 1 | 11
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 3 | 4
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of very severe RSV LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0013, Exact method using binomial distribution; Efficacy = 75.31, 95% CI 2-sided [38.012 to 91.747]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of very severe RSV LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0620, Exact method using binomial distribution; Efficacy = 78.10, 95% CI 2-sided [-5.823 to 97.697]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of very severe RSV LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0060, Exact method using binomial distribution; Efficacy = 91.01, 95% CI 2-sided [38.156 to 99.791]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of very severe RSV LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.9851, Exact method using binomial distribution; Efficacy = 26.01, 95% CI 2-sided [-337.329 to 89.162]

7. Secondary Outcome: Number of Participants With Hospitalization for All-Cause Lower Respiratory Tract Infection Through 151 Days Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with hospitalization for all-cause LRTI through 151 days post-dosing/randomization in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) to Day 151
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 76 | 132
  France: number analyzed (Participants) | 1090 | 1087
  France | 32 | 48
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 35 | 58
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 9 | 26
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 43.62, 95% CI 2-sided [24.677 to 58.057]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0754, Exact method using binomial distribution; Efficacy = 34.78, 95% CI 2-sided [-4.148 to 59.648]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0177, Exact method using binomial distribution; Efficacy = 40.67, 95% CI 2-sided [8.211 to 62.156]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through Day 151 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0046, Exact method using binomial distribution; Efficacy = 66.38, 95% CI 2-sided [25.952 to 86.137]

8. Secondary Outcome: Number of Participants With Immediate Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were either events with the start date and time posterior to the start of the treatment period and up to the end of the treatment period or events with the start date and time prior to the start of the treatment period, whose severity was greater than 1 or missing and stop date is missing or not before the treatment period. Immediate events were recorded to capture medically relevant AEs which occurred within the first 30 minutes after immunization.
Time Frame: Up to 30 minutes post-dosing/randomization on Day 1
Population: The Safety Analysis Set (SafAS) consisted of all participants who received nirsevimab in the study and all randomized participants who were randomized to the no intervention group and did not receive nirsevimab inadvertently. As pre-specified in the protocol and SAP, results are presented by treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4016 | 4018
Participants | 27 | 0

9. Secondary Outcome: Number of Participants With Non-Serious Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were either events with the start date and time posterior to the start of the treatment period and up to the end of the treatment period or events with the start date and time prior to the start of the treatment period, whose severity was greater than 1 or missing and stop date was missing or not before the treatment period.
Time Frame: From dosing/randomization (Day 1) to Day 31
Population: The SafAS consisted of all participants who received nirsevimab in the study and all randomized participants who were randomized to the no intervention group and did not receive nirsevimab inadvertently. As pre-specified in the protocol and SAP, results are presented by treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4016 | 4018
Participants | 1316 | 1265

10. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAEs), Treatment-Emergent Adverse Events of Special Interest (AESIs) and Treatment-Emergent Medically Attended Adverse Events (MAAEs)
Description: AE: untoward medical occurrence in clinical study participant, temporally associated with use of study intervention, whether or not related to it. TEAEs: events with start date/time posterior to start of treatment period(TP) and up to end of TP, or events with start date/time prior to start of TP, whose severity was>1/missing; stop date was missing/not before TP. SAE: AE at any dose resulting in death, persistent or significant disability/incapacity, required inpatient hospitalization/prolongation of existing hospitalization, was life-threatening or congenital anomaly/birth defect or medically important event. MAAE: new onset/worsening of condition that prompted participant or participant's parent/legally acceptable representative to seek unplanned medical advice at physician's office/Emergency Department. AESI: scientific, medical concern specific to Sponsor's study intervention/program for which ongoing monitoring and rapid communication by investigator to Sponsor was appropriate.
Time Frame: From dosing/randomization (Day 1) to Day 366
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4016 | 4018
Participants
  Treatment-emergent SAEs | 262 | 222
  Treatment-emergent AESIs | 11 | 3
  Treatment-emergent MAAEs | 3106 | 3100

11. Secondary Outcome: Number of Participants With Treatment-Related Serious Adverse Event (for United Kingdom Reconsented Participants)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were either events with the start date and time posterior to the start of the treatment period and up to the end of the treatment period or events with the start date and time prior to the start of the treatment period, whose severity was greater than 1 or missing and stop date is missing or not before the treatment period. SAE: AE at any dose resulting in death, persistent or significant disability/incapacity, required inpatient hospitalization/prolongation of existing hospitalization, was life-threatening or congenital anomaly/birth defect or medically important event. A treatment-related TEAE was a TEAE considered by the investigator as related or with unknown/missing relationship to treatment for participants who received nirsevimab on Day 1.
Time Frame: From Day 366 to Day 731
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 1140 | 1084
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Respiratory Syncytial Virus Lower Respiratory Tract Infection Hospitalization Through 181 Days Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with RSV LRTI hospitalization through 181 days post-dosing/randomization in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) to Day 181
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 12 | 68
  France: number analyzed (Participants) | 1090 | 1087
  France | 4 | 28
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 3 | 21
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 5 | 19
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations through Day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 82.72, 95% CI 2-sided [67.826 to 91.490]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations through Day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 86.13, 95% CI 2-sided [60.340 to 96.464]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations through Day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0002, Exact method using binomial distribution; Efficacy = 85.92, 95% CI 2-sided [52.850 to 97.311]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of RSV LRTI hospitalizations through Day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0054, Exact method using binomial distribution; Efficacy = 74.39, 95% CI 2-sided [29.077 to 92.525]

13. Secondary Outcome: Number of Participants With Hospitalization for All-Cause Lower Respiratory Tract Infection Through 181 Days Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with hospitalization for all-cause LRTI through 181 days post-dosing/randomization in France, UK, Germany, and overall is presented.
Time Frame: From dosing/randomization (Day 1) to Day 181
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4038 | 4019
Participants
  Overall | 82 | 138
  France: number analyzed (Participants) | 1090 | 1087
  France | 34 | 49
  United Kingdom: number analyzed (Participants) | 2052 | 2039
  United Kingdom | 38 | 62
  Germany: number analyzed (Participants) | 896 | 893
  Germany | 10 | 27
Statistical Analysis 1: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Overall: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p < 0.0001, Exact method using binomial distribution; Efficacy = 41.89, 95% CI 2-sided [23.073 to 56.333]
Statistical Analysis 2: Comparison: Nirsevimab vs No Intervention; Statistical analysis for France: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.1003, Exact method using binomial distribution; Efficacy = 32.19, 95% CI 2-sided [-7.188 to 57.545]
Statistical Analysis 3: Comparison: Nirsevimab vs No Intervention; Statistical analysis for UK: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0164, Exact method using binomial distribution; Efficacy = 39.83, 95% CI 2-sided [8.449 to 60.911]
Statistical Analysis 4: Comparison: Nirsevimab vs No Intervention; Statistical analysis for Germany: The 2-sided 95% CI for the efficacy was calculated by an exact method assuming a binomial distribution of the number of hospitalizations for all-cause LRTI through day 181 post-dosing/randomization in the nirsevimab group conditional on the total number in both groups accounting for the follow-up time post-dosing/randomization; Test type: Superiority; p = 0.0058, Exact method using binomial distribution; Efficacy = 64.06, 95% CI 2-sided [23.386 to 84.478]

14. Secondary Outcome: Number of Participants With Respiratory Syncytial Virus Lower Respiratory Tract Infection Hospitalization From Days 181 to 366 Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with RSV LRTI hospitalization from Days 181 to 366 post-dosing/randomization (with no RSV LRTI hospitalizations before Day 181) in France, UK, Germany, and overall is presented.
Time Frame: From Day 181 to Day 366
Population: The All Randomized Set consisted of all participants randomly assigned to either the nirsevimab group or the no intervention group. Only participants with data collected are reported. 'Number Analyzed' indicates the number of participants with data collected for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 4026 | 3951
Participants
  Overall | 31 | 28
  France: number analyzed (Participants) | 1086 | 1059
  France | 6 | 5
  United Kingdom: number analyzed (Participants) | 2049 | 2018
  United Kingdom | 20 | 19
  Germany: number analyzed (Participants) | 891 | 874
  Germany | 5 | 4

15. Secondary Outcome: Number of Participants With Hospitalization for All-Cause Lower Respiratory Tract Infection From Days 181 to 366 Post-dosing/Randomization
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with hospitalization for all-cause LRTI from Days 181 to 366 post-dosing/randomization (with no hospitalizations for all-cause LRTI before Day 181) is presented.
Time Frame: From Day 181 to Day 366
Population: The All Randomized Set consisted of all participants randomly assigned to either the nirsevimab group or the no intervention group. Only participants with data collected are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 3956 | 3881
Participants | 68 | 55

16. Secondary Outcome: Number of Participants With Respiratory Syncytial Virus Lower Respiratory Tract Infection Hospitalization From Days 366 to 731 Post-dosing/Randomization (for United Kingdom Reconsented Participants)
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with RSV LRTI hospitalization from Days 366 to 731 post-dosing/randomization (with no RSV LRTI hospitalizations before Day 366) in UK reconsented participants is presented.
Time Frame: From Day 366 to Day 731
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 1132 | 1062
Participants | 7 | 2

17. Secondary Outcome: Number of Participants With Hospitalization for All-Cause Lower Respiratory Tract Infection From Days 366 to 731 Post-dosing/Randomization (for United Kingdom Reconsented Participants)
Description: LRTI included the following common symptoms: clinical finding of rhonchi, rales, crackles, or wheeze; increased respiratory rate at rest (age: <2 months, ≥60 breaths/min; 2 to 6 months, ≥50 breaths/min; >6 months, ≥40 breaths/min), and hypoxemia (in room air: oxygen saturation <95%). Hospitalization was defined as the decision to admit to in-patient care by the treating physician. Number of participants with hospitalization for all-cause LRTI from Days 366 to 731 post-dosing/randomization (with no hospitalizations for all-cause LRTI before Day 366) in UK reconsented participants is presented.
Time Frame: From Day 366 to Day 731
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 1096 | 1025
Participants | 18 | 10

18. Secondary Outcome: Number of Participants With Recurrent Wheeze (for United Kingdom Reconsented Participants)
Description: Wheeze was defined as a physician-diagnosed wheeze or asthma or related ear, nose and throat (ENT)/respiratory symptoms at an office visit or an illness for which the child was prescribed medication to treat an ENT/respiratory condition. Recurrent wheeze event was defined as 2 or more protocol-defined wheeze episodes throughout follow-up period.
Time Frame: From dosing/randomization (Day 1) to Day 731
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab | No Intervention
Number analyzed (Participants) | 928 | 888
Participants | 101 | 96

ADVERSE EVENTS:
Time Frame: SAEs and all-cause mortality were collected from dosing/randomization (Day 1) up to end of follow-up (Day 366 for France, Germany, UK non-reconsented participants and Day 731 for UK reconsented participants). Non-serious AEs were collected from dosing/randomization (Day 1) up to Day 31 as pre-specified in protocol.
Description: Analysis was performed on the SafAS. As pre-specified in the protocol and SAP, results are presented by treatment group. Safety analysis was not planned exclusively for UK reconsented participants, and no separate safety data was collected for this subgroup.
Arm/Group | Nirsevimab | No Intervention
All-Cause Mortality (participants affected / at risk) | 1/4016 | 0/4018
Serious Adverse Events (participants affected / at risk) | 262/4016 | 222/4018
Other Adverse Events (participants affected / at risk) | 324/4016 | 279/4018
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirsevimab (N=4016) | No Intervention (N=4018)
Accidental Exposure To Product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 3 (4) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign Body In Gastrointestinal Tract (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign Body Ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Stoma Prolapse (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Coronavirus Test Positive (Investigations) | 1 (1) | 0 (0)
Human Rhinovirus Test Positive (Investigations) | 0 (0) | 1 (1)
Oxygen Saturation Decreased (Investigations) | 3 (3) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bicuspid Aortic Valve (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Birth Mark (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cataract Congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Choanal Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cleft Palate (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Coarctation Of The Aorta (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital Megacolon (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Craniofacial Deformity (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Factor Viii Deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypospadias (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Kabuki Make-Up Syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pulmonary Sequestration (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Urethral Valves (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Altered State Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (4) | 2 (2)
Febrile Convulsion (Nervous system disorders) | 10 (11) | 10 (12)
Fontanelle Bulging (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 0 (0) | 1 (1)
Infantile Spasms (Nervous system disorders) | 2 (2) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Petit Mal Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 11 (11) | 3 (3)
Seizure Like Phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 2 (2)
Tonic Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive To Stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Eye Disorder (Eye disorders) | 0 (0) | 1 (1)
Eye Movement Disorder (Eye disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 5 (5) | 5 (6)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (2) | 3 (5)
Intestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 2 (2)
Protein-Losing Gastroenteropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 4 (7)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acne Infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Feeding Disorder (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Food Refusal (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight Gain Poor (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Abscess Neck (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus Infection (Infections and infestations) | 2 (2) | 2 (2)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Beta Haemolytic Streptococcal Infection (Infections and infestations) | 1 (1) | 1 (1)
Bullous Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 6 (6) | 8 (8)
Cellulitis Orbital (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus Infection (Infections and infestations) | 6 (6) | 2 (2)
Croup Infectious (Infections and infestations) | 5 (5) | 3 (3)
Cytomegalovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis Infected (Infections and infestations) | 1 (1) | 0 (0)
Dermo-Hypodermitis (Infections and infestations) | 0 (0) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0)
Ear Infection Viral (Infections and infestations) | 1 (1) | 0 (0)
Eczema Herpeticum (Infections and infestations) | 1 (1) | 1 (1)
Eczema Infected (Infections and infestations) | 0 (0) | 2 (2)
Enterovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Gastric Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 11 (12) | 12 (12)
Gastroenteritis Adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Enteroviral (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis Norovirus (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis Rotavirus (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 4 (4) | 2 (2)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 4 (4)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious Mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 8 (8) | 6 (6)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 3 (3)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0)
Lymph Node Abscess (Infections and infestations) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 1 (1) | 2 (2)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Enteroviral (Infections and infestations) | 1 (1) | 1 (1)
Meningitis Neonatal (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Norovirus Infection (Infections and infestations) | 2 (2) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 2 (2) | 1 (1)
Otitis Media Acute (Infections and infestations) | 0 (0) | 2 (2)
Parainfluenzae Virus Infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 10 (12) | 9 (11)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 (1) | 2 (2)
Respiratory Tract Infection Viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 3 (3) | 3 (3)
Roseola (Infections and infestations) | 2 (2) | 0 (0)
Rotavirus Infection (Infections and infestations) | 1 (1) | 2 (2)
Salmonellosis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Staphylococcal Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subglottic Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Suspected Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 7 (7) | 2 (2)
Tonsillitis Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 10 (10) | 9 (9)
Urachal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 7 (7) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Viral Diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 11 (11) | 7 (7)
Viral Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral Rash (Infections and infestations) | 1 (1) | 0 (0)
Viral Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 4 (4)
Cyanosis (Vascular disorders) | 1 (1) | 1 (1)
Kawasaki's Disease (Vascular disorders) | 2 (2) | 1 (1)
Acute Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Allergy To Vaccine (Immune system disorders) | 1 (1) | 0 (0)
Alloimmunisation (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 2 (2)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Food Allergy (Immune system disorders) | 4 (5) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Milk Allergy (Immune system disorders) | 0 (0) | 1 (1)
Crying (General disorders) | 1 (1) | 0 (0)
Electrocution (General disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 1 (1)
Hyperthermia (General disorders) | 2 (2) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 9 (9) | 11 (12)
Breath Holding (Psychiatric disorders) | 1 (1) | 0 (0)
Stereotypy (Psychiatric disorders) | 0 (0) | 1 (1)
Breast Inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular Torsion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Brief Resolved Unexplained Event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (5)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirsevimab (N=4016) | No Intervention (N=4018)
Nasopharyngitis (Infections and infestations) | 324 (345) | 279 (298)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/10/NCT05437510/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT05437510/SAP_001.pdf